CLINICAL TRIAL: NCT02828215
Title: A Prospective Study to Evaluate Swept-Source OCT and Adaptive Optics Imaging of Diseases of the Vitreous, Retina and Choroid
Brief Title: Advanced OCT and Adaptive Optics Imaging in Retinal Disease (The ACAD Study)
Acronym: ACAD
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PATP1022
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Vitreous Diseases; Retinal Diseases; Choroidal Diseases
MeSH Terms: conditions — Retinal Diseases; Choroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Swept-source optical coherence tomography (SS-OCT) — The SD-OCT provides faster images and the ability to scan more of the central retina (macula). SD-OCT simultaneously measures multiple wavelengths of reflected light across a spectrum generating up to 40,000 A-Scans (axially sample points) per second. This allows the generation of 3 dimensional faster based volumetric images of the retina. The Spectralis OCT utilises real-time hardware eye tracking to resample lines scan enhancing the signal to noise ratio by improving the image quality.
  The swept-source OCT (SS-OCT) uses a tuneable laser light source with a longer wavelength of light (typically 1040-1050 nm) that the light source seen in more conventional SD-OCT devices. The tissue penetration and resolution is greater with fast acquisition speeds and longer line scan lengths.
  Other Names: Spectral Domain coherence topography (SD-OCT); Adaptive Optics Scanning light ophthalmoscope (AOSLO)

SUMMARY:
The objectives of this study include using the new technology of SS-OCT (swept source optical coherence tomography) to evaluate morphological abnormalities of the vitreous, retina and choroid and to assess the repeatability of retinal and choroidal thickness measurements in retinal disease using SS-OCT. A secondary objective is to use the new imaging modality of adaptive optics to directly visualize photoreceptor mosaics and microvasculature in eyes with retinal and choroidal disease.

DETAILED DESCRIPTION:
Diseases affecting the vitreous, retina and choroid are among the commonest causes of sight-loss and vision impairment in England and Wales.

These diseases may display a wide range of pathological features including vitreous, retinal and subretinal haemorrhage; macular fluid; choroidal inflammation and choroidal masses.

The retina is a 'window to the brain' and there is increasing evidence that neurodegenerative disorders such as Multiple Sclerosis, Parkinsons Disease and Alzheimers Disease have retinal manifestations which may have prognostic implications, afford earlier diagnosis, and potentially act as surrogate endpoints for treatment trials.

In 2012, a further advance in OCT technology was brought to market with the arrival of the first commercial available swept-source OCT (SS-OCT) device (the Topcon DRI OCT). SS-OCT technology uses a tuneable laser light source with a longer wavelength of light (typically 1040-1050 nm central wavelength) than the light sources seen in more conventional SD-OCT devices. This leads to greater tissue penetration with less backscatter from the RPE, producing images of the choroid with greater resolution with fast image acquisition speeds (100,000 A scans/s) and longer line scan lengths. The ability to take rapid scans with the only commercially available SS-OCT device (the DRI, Tocon Inc. Paramus, NY, USA) also enhances image quality by line scan averaging capability.

The high axial resolution of OCT allows discrimination of the distinct retinal layers that are affected differentially in different diseases. More direct visualisation of the photoreceptor layer is afforded by use of an Adaptive Optics Scanning Light Ophthalmoscope (AOSLO), which provides excellent lateral resolution and allows direct visualisation of the cone and rod photoreceptor mosaics in vivo by correcting for ocular aberrations and resulting in a lateral comparable with histopathological sections.

In this study AO images will be correlated with SD- and SS-OCT and used to comprehensively assess the integrity of the photoreceptor mosaic. Furthermore AO and OCT will be used to measure nerve fibre layer loss and optic disc changes if relevant to the disease.

The imaging modalities used in this study will be spectral domain optical coherence topography (SD-OCT), swept source optical coherence tomography (SS-OCT), and adaptive optics scanning light ophthalmoscope (AOSLO)

The study will examine 300 patients (up to 600 eyes) in a single visit with a further Adaptive Optics (AO) imaging taken in a subset of patients (up to 200).

Patients in whom AO imaging was possible from a technical perspective will be invited back for further imaging after 6-12 months (at a standard NHS follow up visit) to probe longitudinal changes.

An examiner will scan the participants study eye(s) on the same day on each of the 3 imaging modalities SD-OCT, SS-OCT and AOSLO.

Finally a questionnaire will be used to explore whether participants preferred one OCT imaging modality over the other (SS-OCT vs SD-OCT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients attending Moorfields Eye Hospital with a diagnosis of diseases of the vitreous, retina or choroid in at least one eye including but not restricted to:

   1. Vitritis
   2. Vitreomacular interface abnormalities including macular hole
   3. Age-related macular degeneration
   4. Diabetic macular oedema and retinopathy
   5. Other causes of macular oedema
   6. Inherited retinal dystrophies
   7. Inherited macular dystrophies
   8. Posterior Uveitis (infectious and non-infectious)
   9. Retinal nerve fibre layer loss (eg due to glaucoma)
2. Patients with neurodegenerative diseases such as multiple sclerosis for which there is previous literature identifying retinal/choroidal abnormalities referred by Consultant Neurologists within UCL Partners
3. Male or female aged 18 years old or over.
4. Ability to understand nature/purpose of study and to provide informed consent
5. Ability to undergoing imaging
6. Ability to follow instructions and complete study

Exclusion Criteria:

1. History of previous significant ocular trauma
2. Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule or other study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending Moorfields Eye Hospital with a diagnosis of diseases of the vitreous, retina or choroid in at least one eye
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
3 repeated measurements of choroid + retinal thickness using SD-OCT and SS-OCT and optic nerve head imaging | 3 years

SECONDARY OUTCOMES:
Percentage concordance and Kappa statistics of detection of morphological abnormalities in widefield OCT and conventional filed OCT (Spectralis OCT) | 3 years
Repeated measures of photoreceptor mosaic integrity and microsvasculature (subset of patients only) at 2 visits | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Patel, MBBChir MA FRCOphth MD(Res), Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- NIHR Clinical Research Facility - Moorfileds Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanumunthadu D, Keane PA, Balaskas K, Dubis AM, Kalitzeos A, Michaelides M, Patel PJ. Agreement Between Spectral-Domain and Swept-Source Optical Coherence Tomography Retinal Thickness Measurements in Macular and Retinal Disease. Ophthalmol Ther. 2021 Dec;10(4):913-922. doi: 10.1007/s40123-021-00377-8. Epub 2021 Jul 29. PMID 34324166